CLINICAL TRIAL: NCT05812950
Title: Clinical and Cost-effectiveness of Group Schema Therapy for Complex Eating Disorders: the GST-EAT Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Utrecht University (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); GGNet Amarum (Unknown); GGZ Breburg (Other); Accare (Other); Co-eur (Unknown); GGZ Friesland (Other); University of Groningen (Other)
Responsible Party: Principal Investigator, Jeffrey Roelofs, Principal investigator J. Roelofs, PhD, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL80491.068.22; 60-63600-98-1131 (Registry Identifier: ZonMw)
Record Dates: First submitted 2023-03-04; First posted 2023-04-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Anorexia Nervosa; Atypical Anorexia Nervosa (Other Specified Eating Disorder); Bulimia Nervosa; Atypical Bulimia Nervosa (Other Specified Eating Disorder)
Keywords: CBT-E; Group Schema Therapy; Eating disorders; Effectiveness
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: All participants start with CBT-E phase 1 and 2. If not improved enough with regard to eating disorder symptoms (following EDE-Q pre- and post measure comparison) in the first phase, they will be included in the RCT. When included they will be randomly assigned to either the CBT-E continuation condition or the GST condition.
Who Masked: Outcomes Assessor
Masking Description: Once data collection is complete, the data will be blinded by one of the principal investigators. This allows for blinded analysis by the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Schema Therapy for eating disorders (GST) (Experimental): GST starts with 5 individual sessions for introducing the ST model, placing the ED symptoms and behaviors in the context of coping modes, and organizing these in a mode map conceptualization. Thereafter there are 26 weekly group sessions of ST for EDs, supplemented with 8 optional individual ST sessions, and a psycho-education webinar for relatives. The sessions focus on recognizing and changing personal coping modes and underlying early maladaptive schemas, and developing and strengthening the healthy adult mode. GST combines interpersonal, experiential, cognitive and behavioral elements in a unified ST approach (Farrell et al., 2014). Although not at the core of GST, addressing the physiological aspects of the ED (weight care and (restrictive) eating) is necessary and therefore also incorporated in the protocol.
  Note that the participants in this condition have followed phase 1 and 2 of CBT-E before starting the GST, as following these phases is required to be included in the RCT.
  Interventions: Behavioral: GST
- Cognitive Behavioral Therapy-Enhanced (CBT-E) (TAU) (Active Comparator): This transdiagnostic ED treatment (current standard of care/treatment of choice) consists of 20-40 individual therapy sessions, based on the transdiagnostic CBT model of EDs. CBT-E consists of four phases. In phase one, the patient creates a personal case formulation, and the focus is on psycho-education on maintaining factors and at starting well with monitoring eating behaviours and establishing a regular eating pattern. In phase two, the first phase is evaluated and a treatment plan is made. In phase three, the main mechanisms that are thought to maintain the patient's ED (over-evaluation of shape, weight, and eating, dietary restraint or restriction, being underweight, and event- or mood-triggered changes in eating behaviour), are targeted, and a relapse plan is created. Phase four focuses on evaluating the progress so far and maintaining the changes that have been obtained (Fairburn et al., 2009).
  Interventions: Behavioral: CBT-E

INTERVENTIONS:
Behavioral: GST — Outpatient eating disorder treatment (5 individual pre-group sessions followed by 26 weekly group sessions + 8 optional individual sessions)
  Arms: Group Schema Therapy for eating disorders (GST)
Behavioral: CBT-E — Outpatient eating disorder treatment (20-40 weekly individual sessions)
  Arms: Cognitive Behavioral Therapy-Enhanced (CBT-E) (TAU)

SUMMARY:
Amongst psychiatric illnesses, eating disorders (EDs) are notoriously difficult to treat and have a high mortality rate. The average duration of an ED is 6 years and for a majority of ED patients, the disorder will become chronic. Comorbid personality pathology such as negative core beliefs and early maladaptive schemas (EMS) are strongly related to ED severity and chronicity. Enhanced cognitive-behavioural therapy for eating disorders (CBT-E) is used as the first line transdiagnostic treatment for EDs. However, CBT-E is mainly symptom-focused and does not tap into these underlying core beliefs and EMS.

Given the limited treatment effects of existing ED treatments, and the importance of comorbid personality pathology, there is an urgent need to examine more effective treatments for EDs. Group-schematherapy (GST) overcomes the limitations of CBT-E and preliminary results for treatment-resistant EDs are promising. However, robust evidence regarding the clinical and cost-effectiveness of GST for patients that do not benefit from CBT-E is not yet available. The central aim of this project is to investigate the clinical and cost-effectiveness of GST for EDs in patients with comorbid personality pathology, who do not show a clinically significant response in the first phase of CBT-E. This is relevant and important as studies examining the effectiveness of GST for EDs are scarce. This project is a joint research initiative of three academic centers (Dutch Universities), four large nation-wide mental health organizations, and two foundations for client empowerment and participation. Eligible patients will be randomized to either GST or continuation of their CBT-E treatment after failing to show a significant treatment response in the first phase of CBT-E. Based on encouraging findings from previous studies and our own pilot data, a statistically and clinically significant better outcome in terms of ED symptoms, negative core beliefs, EMS, schema modes, and quality of life is expected in the GST group compared to the CBT-E group. GST is also expected to be more cost-effective compared to CBT-E as GST may in the long run prevent chronicity in terms of long treatment trajectories and delayed recovery. Finally, with the proviso of good results for GST, we will disseminate and implement GST in the standard of care for EDs. This project thereby has great potential to improve clinical and cost-effectiveness of treatment for chronic EDs.

ELIGIBILITY:
Inclusion Criteria:

* 1) age > 16 years;
* 2) a DSM-5 diagnosis of anorexia nervosa, bulimia nervosa, or other specified ED (atypical anorexia nervosa or bulimia nervosa with a low frequency or limited duration).

Exclusion Criteria:

* 1) not being able to speak and read the Dutch language;
* 2) being in an acute psychotic mental health state at the start of the study;
* 3) being diagnosed with an autism spectrum disorder;
* 4) having an IQ below 80, as determined with a validated instrument;
* 5) showing an early response after phase 1 of CBT-E.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Eating Disorder Examination Questionnaire (EDE-Q) score | Baseline (Before start CBT-E), 4 weeks (8 sessions CBT-E), end of treatment (up to 39 weeks after randomization), and 6 and 12 months after end of treatment
  Eating pathology will be measured with the Eating Disorder Examination Questionnaire (EDE-Q). Fairburn & Beglin, 2008). This self-report measure is the most commonly used routine outcome measure in ED facilities in the Netherlands to measure the severity of the ED.

SECONDARY OUTCOMES:
Childhood Trauma Questionnaire-Short Form (CTQ-SF) | Baseline (Before start CBT-E)
  This questionnaire consists of 28 questions measuring physical abuse, emotional abuse, sexual abuse, physical neglect and emotional neglect during childhood.
Change in Young Schema Questionnaire Short Form version 3 3 (YSQ-S3) score | Baseline (Before start CBT-E), end of treatment (up to 39 weeks after randomization), and 6 and 12 months after end of treatment
  The YSQ-S3 will be used to measure 18 early maladaptive schemas and is a valid instrument for the assessment of early maladaptive schemas in clinical and research settings.
Change in Schema Mode Inventory for Eating Disorders (SMI-ED) score | 4 weeks (8 sessions CBT-E), end of treatment (up to 39 weeks after randomization), and 6 and 12 months after end of treatment
  The SMI-ED will be used to assess schema modes that are relevant in patients with an eating disorder. It measures 5 maladaptive child modes, 2 maladaptive internalized/introject modes, 7 maladaptive coping modes, and 2 healthy factors.
Change in Brief Symptom Inventory (BSI) score | 4 weeks (8 sessions CBT-E), end of treatment (up to 39 weeks after randomization), and 6 and 12 months after end of treatment
  The BSI will be used to assess general psychological and physical symptoms
Change in Eating Disorder Quality of Life (EDQoL) score | 4 weeks (8 sessions CBT-E), end of treatment (up to 39 weeks after randomization), and 6 and 12 months after end of treatment
  Quality of life will be assessed using the EDQoL
Clinical Perfectionism Questionnaire (CPQ) | Baseline (Before start CBT-E)
  The CPQ will be used to assess clinical perfectionism. This questionnaire consists of 12 items that measure the level of self-evaluation based on striving towards extremely high personal standards despite adverse consequences.
Session Rating Scale (SRS) | up to 39 weeks
  Therapeutic alliance will be evaluated in each session using the patient-rated SRS, which is a short (four items) measure.
Quality of life and achievement personalized treatment goals | End of treatment (up to 39 weeks after randomization)
  A qualitative interview (to be developed)
Treatment Inventory of Costs in Patients with psychiatric disorders (TiC-P) | 4 weeks (8 sessions CBT-E), end of treatment (up to 39 weeks after randomization), and 6 and 12 months after end of treatment
  Patient-reported productivity losses and multiple dimensions of healthcare resource consumption will be measured, using the validated TIC-P questionnaire. This questionnaire has been tested extensively for patients with a psychiatric disorder, using a recall period of three months. Using various unit prices in healthcare, both productivity losses and healthcare resource consumption will be valued monetarily in order to estimate the actual costs for the CBT-E arm and the GST arm within a closed time frame (Bouwmans et al., 2013).
Change in Quality-adjusted life years score | 4 weeks (8 sessions CBT-E), end of treatment (up to 39 weeks after randomization), and 6 and 12 months after end of treatment
  Five dimensions of quality of life will be measured, using the EQ-5D-5L questionnaire: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Participants will be asked to rank the extent to which they feel satisfied about these five dimensions on a 5-point Likert scale. Then they will be asked to rank their current health state, using a 0-100 VAS analog scale. Final utility scores from both the CBT-E arm and the GST arm on all dimensions of this questionnaire will be converted into a single health utility measure: Quality-adjusted life years or QALYs (Feng et al., 2021).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Roelofs, Principal Investigator — Maastricht University
Locations (7):
- Netherlands (7):
  - GGz Breburg, Breda
  - Accare, Groningen
  - GGZ Friesland, Leeuwarden
  - GGNet Amarum, Nijmegen
  - GGz Breburg, Tilburg
  - Co-eur, Utrecht
  - GGNet Amarum, Warnsveld

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mares SHW, Roelofs J, Zinzen J, Beatse M, Elgersma HJ, Drost RMWA, Evers SMAA, Elburg AAV. Clinical effectiveness, cost-effectiveness and process evaluation of group schema therapy for eating disorders: study protocol for a multicenter randomized controlled trial. BMC Psychol. 2024 Mar 4;12(1):123. doi: 10.1186/s40359-024-01624-w. PMID 38439092